CLINICAL TRIAL: NCT00002905
Title: PROSPECTIVE NON-RANDOMIZED STUDY WITH CHEMOTHERAPY FOR RELAPSED OR REFRACTORY HIV-RELATED NON-HODGKIN'S LYMPHOMA: VMP REGIMEN FOR RELAPSED PATIENTS, CDE REGIMEN FOR REFRACTORY PATIENTS
Brief Title: Combination Chemotherapy in Treating Patients With HIV-Related Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065256; ITA-GICAT-C-941202-3; EU-96059
Record Dates: First submitted 1999-11-01; First posted 2004-06-09 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2011-09

CONDITIONS: Lymphoma
Keywords: AIDS-related peripheral/systemic lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Cyclophosphamide; Didanosine; Doxorubicin; Etoposide; Mitoxantrone; Prednimustine; Zidovudine

INTERVENTIONS:
Drug: cyclophosphamide
Drug: didanosine
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: mitoxantrone hydrochloride
Drug: prednimustine
Drug: zidovudine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients with HIV-related non-Hodgkin's lymphoma that has relapsed or has not responded to chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the response rate and duration of response to etoposide, mitoxantrone, and prednimustine in patients with relapsed HIV-associated non-Hodgkin's lymphoma (NHL). II. Evaluate the response rate and duration of response to cyclophosphamide, doxorubicin, and etoposide in patients with refractory HIV-associated NHL. III. Assess the toxic effects of these regimens in these patients.

OUTLINE: Patients with relapsed non-Hodgkin's lymphoma (NHL) receive oral etoposide and prednimustine on days 1-5 and intravenous mitoxantrone on day 1 every 3 weeks. Patients with refractory NHL receive cyclophosphamide, doxorubicin, and etoposide as a continuous infusion over 4 days every 4 weeks. All patients receive concomitant antiretroviral therapy with zidovudine or didanosine. G-CSF is given for hematologic support as indicated. All patients are evaluated for response after 2 courses of chemotherapy. Patients with a complete response (CR) receive 2 additional courses. Patients with a stable or partial response receive 2 additional courses and are re-evaluated; those with a CR receive 2 more courses, while those with a stable or partial response are treated off study at the physician's discretion. Patients with progressive disease are removed from study.

PROJECTED ACCRUAL: 15-20 patients will be treated on each regimen.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven non-Hodgkin's lymphoma at first presentation No documented CNS involvement (i.e., primary CNS or meningeal lymphoma) Positive serologic test for HIV antibodies required No opportunistic infection unless effectively treated Disease relapsed, refractory, or unresponsive to first-line chemotherapy No more than 1 prior combination chemotherapy regimen Chemotherapy consisted of cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) or a CHOP-like regimen, ACVBP, or other similar regimen

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-3 Life expectancy: At least 1 month Hematopoietic: Not specified Hepatic: Bilirubin less than 5 times normal OR Transaminases less than 5 times normal Renal: Creatinine less than 2 mg/dL

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 1995-06

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Tirelli, MD, Study Chair — Centro di Riferimento Oncologico - Aviano
Locations (1):
- Centro di Riferimento Oncologico - Aviano, Aviano, Italy